CLINICAL TRIAL: NCT01386866
Title: An Open-label, Single Dose Study of the Mass Balance and Metabolic Disposition of Orally Administered [14C]-Labelled AMG 706 (Motesanib) Followed by Extended Treatment With Motesanib in Patients With Advanced Solid Tumors
Brief Title: Single Dose Study of [14C]-Labelled AMG 706 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20080639
Record Dates: First submitted 2011-04-14; First posted 2011-07-01 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Advanced Solid Tumors
Keywords: AMG 706; Motesanib; Amgen; Phase 1
MeSH Terms: interventions — motesanib diphosphate

ARMS (1):
- A (Experimental)
  Interventions: Drug: AMG 706

INTERVENTIONS:
Drug: AMG 706 — Single oral dose of 125 mg AMG 706 (motesanib) containing 100 μCi of [14C]-AMG 706 followed by option to continue onto a treatment extension phase for potential treatment benefit. Subjects will be administered motesanib 125 mg (5 x 25 mg tablets) on a daily basis until subjects experience a dose-limiting toxicity (DLT), an unacceptable AE, disease progression, or voluntary withdrawal.

SUMMARY:
In order for a tumour to grow and spread to other parts of the body, it needs to have a blood supply. Certain proteins in the body, called cytokines or growth factors, have been shown to cause the growth of new blood vessels that supply tumours and therefore help the tumour to grow and spread. Motesanib (AMG 706) prevents these proteins from working, and may help to prevent the growth of tumours.

In the first part of this study, we will look at the way your body absorbs this drug into your blood, how your body changes and breaks down the drug, and then how the drug leaves your body in your urine and faeces.

In order to provide potential treatment benefit for the subjects who participated in the first part of the study, the second part of the study will allow subjects to continue on motesanib (AMG 706) treatment. The estimated length of this part of the study is unknown, and dependent on how subjects respond to motesanib (AMG 706).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a pathologically documented and definitively diagnosed advanced solid tumor(excluding tumors that may significantly interfere with the absorption, metabolism, or excretion of the test article, such as primary or metastatic liver tumor with approximately >50% of liver tissue involvement) that is refractory to standard treatment or for which no curative therapy is available
* Eastern Cooperative Oncology Group performance status of 0-1
* Man or woman (male or female), age > 18 years
* Ability to understand and sign an Independent Ethics Committee (IEC) Approved informed
* Subjects must also fulfil Haematological, Renal, Hepatic and Coagulation criteria (not listed)

Exclusion Criteria:

* Acute disease state (e.g. nausea, vomiting, fever, diarrhea) within 7 days of Day 1
* History of documented arterial or venous thrombosis within 1 year of Day 1
* History of bleeding diathesis or bleeding within 14 days of Day 1, or hypercoagulopathy syndrome
* History of life-threatening ventricular arrhythmia (e.g. sustained ventricular tachycardia)
* History of pulmonary hemorrhage or gross hemoptysis (1/2 teaspoon of bright red blood or more) within 6 months of Day 1
* Central nervous system metastases (exception: subjects with treated, asymptomatic central nervous system metastases, those who have been clinically stable in the judgment of the investigator and off steroids for at least 30 days before Day 1 are eligible)
* Subjects with non-small cell lung cancer (NSCLC)
* Subjects with head and neck cancer
* Subjects with ovarian cancer
* Subjects with large central (located adjacent to or within the hilum or mediastinum) tumor lesions ≥ 3 cm, regardless of histology
* Uncontrolled hypertension: average systolic blood pressure > 150 mm Hg or average diastolic blood pressure > 90 mm Hg (average blood pressure of the three separate blood pressure values measured within 10 minutes during screening)
* Systemic chemotherapy within 28 days of Day 1
* Radiotherapy within 28 days of Day 1 or within 14 days of Day 1 for peripheral lesions
* Experimental or approved antibody therapy within 6 weeks before Day 1
* Concurrent or prior (within 4 weeks prior to Day 1 of 5 half-lives of the medication which ever is longer) treatment with potent CYP3A inducers, including but not limited to : phenytoin, carbamazepine, rifampicin, phenobarbital and St John's Wort
* Concurrent or prior (within 2 weeks prior to Day 1 or 5 half-lives of the medication which ever is longer) treatment with potent CYP3A inhibitors, including but not limited to: ketoconazole, itraconazole, fluconazole, clarithromycin, erythromycin, cyclosporine, tacrolimus, nefazodone and/or HIV protease inhibitors
* Concurrent or prior (within 2 weeks prior to Day 1) consumption of grapefruit (i.e. whole fruit or fruit juice)
* Subjects who as a result of gastrointestinal surgeries (including cholecystectomy) or a medical condition (e.g. constipation, cholecystitis / cholelithiasis) that will significantly alter the absorption, metabolism or excretion of motesanib.
* Subjects with irregular bowel habits (more than 3/day or less than 1 every 2 days).
* Subjects who will not refrain from taking herbal/ complementary therapies (which have the potential to alter the absorption, metabolism, or excretion of the [14C]-AMG 706) for 7 days before first dosing, and for the duration of the ADME part of the study.
* Concurrent immune modulators such as cyclosporine and tacrolimus
* Any anti-coagulation therapy within 7 days prior to Day 1
* Subjects whose occupation requires exposure to radiation or monitoring for radiation exposure
* Clinically significant cardiac disease within 12 months of study Day 1, including myocardial infarction, unstable angina, Grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or ongoing arrhythmias requiring medication
* Major surgery (that which requires general anesthesia) within 28 days or minor surgery within 14 days of Day 1
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures
* History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with study participation or investigational product administration or may interfere with the interpretation of the study results
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection or any co-morbid disease that would increase risk of toxicity
* Any subject not consenting to use adequate contraceptive precautions (eg, hormonal, barrier or abstinence) during the course of the study and for 6 months after the last treatment
* Female subjects who have a positive pregnancy test at screening or on Day-1
* Female subjects who are breastfeeding or plan to breastfeed during the study or within 6 months after the last administration of the investigational product
* Participation in a therapeutic clinical trial within 30 days of Day1
* Subject is unwilling or unable to comply with the study requirements
* Subject has a known sensitivity to any of the products to be administered over the course of the study (e.g. known hypersensitivity to study medication motesanib)
* Subjects with a history of gall bladder and bile duct disease
* Subjects with Gilberts syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Profile and identification of metabolites of [14C]-AMG 706 in plasma, urine, and faeces
Pharmacokinetics of total radioactivity in plasma and whole blood
The mass balance of [14C]-AMG 706 (as the percentage of the dose administered) in urine and faeces

SECONDARY OUTCOMES:
• Measure the area under the plasma concentration curve versus time of AMG 706, as well as determine half-life and time of maximum concentration of AMG 706.
The subject incidences of serious adverse events, adverse events, and clinically significant changes in vital signs and clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com